CLINICAL TRIAL: NCT06104371
Title: Axillary Lymph Node Identification Before Neoadjuvant Chemotherapy Using Magtrace, (Superparamagnetic Iron Oxide Nanoparticles, SPIO) and Magseed, in Clinically Node Negative and Node Positive Patients. SentiNeo 2.0
Brief Title: Lymph Node Identification Using Magtrace and Magseed Before Chemotherapy
Acronym: SentiNeo2
Status: Not yet recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Uppsala University (Other); Region Västmanland (Other); University Hospital, Linkoeping (Other); Baylor College of Medicine (Other); The University of Hong Kong-Shenzhen Hospital (Other); Royal Marsden NHS Foundation Trust (Other); University of Athens (Other); University College Dublin (Other)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, professor, Sahlgrenska University Hospital
Other Study IDs: SUGBG-2023002
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: sentinel lymph node detection; neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Node negative: Clinically node negative before neoadjuvant chemotherapy
  Interventions: Device: Magtrace
- Node positive: Clinically node positive before neoadjuvant chemotherapy
  Interventions: Device: Magtrace

INTERVENTIONS:
Device: Magtrace — Sentinel lymph node tracer and metastatic lymph node clip
  Other Names: Magseed

SUMMARY:
Magnetic tracer injected before preoperative chemotherapy in breast cancer patients for sentinel lymph node detection. Also, magnetic tracer in combination with magnetic clip for index node identification.

DETAILED DESCRIPTION:
This is an interventional single arm study. The aim is to see if sentinel lymph nodes marked with a magnetic tracer injected before preoperative chemotherapy can be detected at surgery three to six moths later. The investigators also want to see if they can find the same nodes with a tracer injected before chemotherapy as with a tracer injected after chemotherapy. The hypothesis is that the chemotherapy might affect the lymph drainage and the nodes marked before the chemotherapy are the true sentinel lymph nodes.

Furthermore, in patients with known lymph node metastases before chemotherapy one metastasis is marked with a magnetic clip before the chemotherapy. This is a well known method but it has not been done in combination with the magnetic tracer. We will show that this is feasible.

All patients included in the study will receive their treatments according to the current standard national guidelines as both the magnetic tracer and the routinely used radioactive tracer are used in parallel. The magnetic clip is also used at several sites in Sweden today.

ELIGIBILITY:
Inclusion criteria:

* Patients 18 years of age or older.
* Patients with breast cancer planned to undergo NACT with

  * planned sentinel lymph node dissection (SLND), or
  * targeted axillary lymph node dissection (TAD), in conjunction with the
* breast surgery after NACT.

Exclusion Criteria:

* Intolerance / hypersensitivity to iron or dextran compounds or SPIO.
* Patients who are required to undergo MRI to evaluate tumour response.
* Pregnancy or breast feedin.g
* Patients with an iron overload disease.
* Patient deprived of liberty or under guardianship.
* Inability to understand given information and give informed consent or undergo study procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients planned for preoperative chemotherapy before breast surgery.
Sampling Method: Non-Probability Sample
Enrollment: 459 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Sentinel lymph node detection rate | Perioperatively
  per patient

SECONDARY OUTCOMES:
Number of sentinel lymph nodes detected per tracer | Perioperatively
  per node
Concordance of nodes per tracer | Perioperatively
  Ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
ON request. Pseudoanonymised data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 months